CLINICAL TRIAL: NCT05202574
Title: Comparing the Effects of Ondansetron Versus Dexamethasone on the Incidence of Post-dural Puncture Headache (PDPH) , Nausea and Vomiting After Spinal Anaesthesia of Parturients Undergoing Caesarean Section
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Mina Maher, Lecturer of anesthesia and ICU, Minia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 278-7/2019
Record Dates: First submitted 2022-01-09; First posted 2022-01-21 (Actual); Last update posted 2022-01-21 (Actual); Status verified 2022-01

CONDITIONS: Post-Dural Puncture Headache
MeSH Terms: conditions — Post-Dural Puncture Headache | interventions — Infusion Pumps

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- dexamethasone (Active Comparator)
  Interventions: Drug: Intravenous drug
- ondanestrone (Active Comparator)
  Interventions: Drug: Intravenous drug
- control group (Placebo Comparator)
  Interventions: Drug: Intravenous drug

INTERVENTIONS:
Drug: Intravenous drug — intravenous drug injection

SUMMARY:
Comparing dexamethasone and ondanestrone injection in ncidence of postdural puncture headache and post-partum nausea and vomiting

ELIGIBILITY:
Inclusion Criteria:

* A total of one hundred and fifty parturients in child bearing period (20-40 years), with BMI of 23-27, and ASA physical status II, who were candidate for elective caesarean section, were enrolled in this prospective randomized study.

Exclusion criteria

Exclusion Criteria:

1 - Lady refusal to participate. 2. All pregnant women candidate for emergency caesarean section elligible for general anaesthesia (GA).

3.presence of any contraindications of dexamethasone (as DM and uncontrolled infection ) or any contraindication of ondansetron (as prolonged QT interval 6. Presence of cardiac, respiratory, hepatic, renal and mental diseases. 7. Coagulopathy, or any contraindication to spinal anaesthesia. 8. Presence of complicated pregnancies (such as pregnancy induced hypertension, placenta previa or eclmpsia).

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-02-01 (Estimated); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
incidence of post-dural puncture hedache | 24 hours post-partum

SECONDARY OUTCOMES:
incidence of post-partum nausea and vomiting | 24 hours post-partum

CONTACTS AND LOCATIONS:
Locations (1):
- Mina Raouf, ALMinya, Minya Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided